CLINICAL TRIAL: NCT04523194
Title: Massachusetts General Hospital and Tsuchiura Kyodo General Hospital Coronary Imaging Collaboration
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Tsuchiura Kyodo General Hospital (Other)
Responsible Party: Principal Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2020P002458
Record Dates: First submitted 2020-08-14; First posted 2020-08-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Coronary Syndrome: Patients diagnosed with acute coronary syndrome.
  Interventions: Other: Optical Coherence Tomography (OCT) and Computed Tomography Angiography (CTA)
- Stable Angina: Patients diagnosed with stable angina.
  Interventions: Other: Optical Coherence Tomography (OCT) and Computed Tomography Angiography (CTA)

INTERVENTIONS:
Other: Optical Coherence Tomography (OCT) and Computed Tomography Angiography (CTA) — Subjects underwent CTA, then OCT during cardiac catheterization as part of their standard clinical care.

SUMMARY:
The purpose of this collaboration is to establish a multi-modality image database including coronary angiograms, optical coherence tomography (OCT), computed tomography angiograms (CTA) and cardiac magnetic resonance imaging (CMR) for future studies. The main goal of this collaboration is to create a resource to promote further understanding of the pathobiology of atherosclerosis through image analysis.

DETAILED DESCRIPTION:
The purpose of this collaboration is to establish a multi-modality image database including coronary angiograms, optical coherence tomography (OCT), computed tomography angiograms (CTA) and cardiac magnetic resonance imaging (CMR) for future studies. About one thousand patients who underwent coronary angiography with OCT and had a CTA prior to catheterization at Tsuchiura Kyodo General Hospital (TKGH) in Japan, will be included. A subset of these patients also had CMR. The main goal of this collaboration is to create a resource to promote further understanding of the pathobiology of atherosclerosis through image analysis.

ELIGIBILITY:
Inclusion Criteria:

* Had CTA prior to cardiac catheterization and then OCT during catheterization

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who underwent CTA prior to cardiac catheterization, and OCT during catheterization were included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 1 Year
  MACE

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Tsuchiura Kyodo General Hospital, Tsuchiura, Japan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD for this observational study.

REFERENCES:
- [Derived] Kinoshita D, Suzuki K, Fujimoto D, Niida T, Minami Y, Dey D, Lee H, McNulty I, Ako J, Ferencik M, Kakuta T, Jang IK. High-risk plaque features and perivascular inflammation. J Cardiovasc Comput Tomogr. 2025 May-Jun;19(3):299-305. doi: 10.1016/j.jcct.2025.01.010. Epub 2025 Feb 7. PMID 39922771
- [Derived] Fujimoto D, Usui E, Vergallo R, Kinoshita D, Suzuki K, Niida T, Covani M, McNulty I, Lee H, Otake H, Shite J, Ferencik M, Dey D, Kakuta T, Jang IK. Relationship Between Coronary Artery Calcium Score and Vulnerability of Culprit Plaque Assessed by OCT in Patients With Established Coronary Artery Disease. Circ Cardiovasc Imaging. 2025 Jan;18(1):e017099. doi: 10.1161/CIRCIMAGING.124.017099. Epub 2024 Dec 20. PMID 39704053
- [Derived] Niida T, Usui E, Suzuki K, Kinoshita D, Yuki H, Fujimoto D, Covani M, Dey D, Lee H, McNulty I, Ferencik M, Yonetsu T, Kakuta T, Jang IK. Differences in total plaque burden between plaque rupture and plaque erosion: A combined computed tomography angiography and optical coherence tomography study. J Cardiovasc Comput Tomogr. 2024 Nov-Dec;18(6):568-574. doi: 10.1016/j.jcct.2024.09.007. Epub 2024 Sep 24. PMID 39322513
- [Derived] Kinoshita D, Suzuki K, Fujimoto D, Niida T, Usui E, Minami Y, Dey D, Lee H, McNulty I, Ako J, Ferencik M, Kakuta T, Jang IK. Relationship between plaque burden and plaque vulnerability: Acute coronary syndromes versus chronic coronary syndrome. J Cardiovasc Comput Tomogr. 2024 Nov-Dec;18(6):559-566. doi: 10.1016/j.jcct.2024.09.002. Epub 2024 Sep 14. PMID 39278792
- [Derived] Fujimoto D, Kinoshita D, Suzuki K, Niida T, Yuki H, McNulty I, Lee H, Otake H, Shite J, Ferencik M, Dey D, Kakuta T, Jang IK. Relationship Between Calcified Plaque Burden, Vascular Inflammation, and Plaque Vulnerability in Patients With Coronary Atherosclerosis. JACC Cardiovasc Imaging. 2024 Oct;17(10):1214-1224. doi: 10.1016/j.jcmg.2024.07.013. Epub 2024 Sep 4. PMID 39243232
- [Derived] Yuki H, Sundt TM, Niida T, Suzuki K, Kinoshita D, Fujimoto D, Dey D, Lee H, McNulty I, Naganuma T, Nakamura S, Usui E, Kakuta T, Jang IK. Level of Perivascular Inflammation Is Significantly Lower Around the Left Internal Mammary Artery Than Around Native Coronary Arteries. J Am Heart Assoc. 2024 Jun 18;13(12):e033224. doi: 10.1161/JAHA.123.033224. Epub 2024 Jun 15. PMID 38879462
- [Derived] Suzuki K, Kinoshita D, Niida T, Yuki H, Fujimoto D, Dey D, Lee H, McNulty I, Takano M, Mizuno K, Ferencik M, Kakuta T, Jang IK. Computed Tomography Angiography Characteristics of Thin-Cap Fibroatheroma in Patients With Diabetes. J Am Heart Assoc. 2024 May 21;13(10):e033639. doi: 10.1161/JAHA.123.033639. Epub 2024 May 14. PMID 38742509
- [Derived] Niida T, Kinoshita D, Suzuki K, Yuki H, Fujimoto D, Dey D, Lee H, McNulty I, Ferencik M, Yonetsu T, Kakuta T, Jang IK. Layered plaque is associated with high levels of vascular inflammation and vulnerability in patients with stable angina pectoris. J Thromb Thrombolysis. 2024 Aug;57(6):880-887. doi: 10.1007/s11239-024-02982-3. Epub 2024 Apr 22. PMID 38649561
- [Derived] Kinoshita D, Suzuki K, Yuki H, Niida T, Fujimoto D, Minami Y, Dey D, Lee H, McNulty I, Ako J, Ferencik M, Kakuta T, Jang IK. Sex-Specific Association Between Perivascular Inflammation and Plaque Vulnerability. Circ Cardiovasc Imaging. 2024 Feb;17(2):e016178. doi: 10.1161/CIRCIMAGING.123.016178. Epub 2024 Feb 20. PMID 38377234
- [Derived] Suzuki K, Kinoshita D, Yuki H, Niida T, Sugiyama T, Yonetsu T, Araki M, Nakajima A, Seegers LM, Dey D, Lee H, McNulty I, Takano M, Kakuta T, Mizuno K, Jang IK. Higher Noncalcified Plaque Volume Is Associated With Increased Plaque Vulnerability and Vascular Inflammation. Circ Cardiovasc Imaging. 2024 Jan;17(1):e015769. doi: 10.1161/CIRCIMAGING.123.015769. Epub 2024 Jan 11. PMID 38205654
- [Derived] Park S, Yuki H, Niida T, Suzuki K, Kinoshita D, McNulty I, Broersen A, Dijkstra J, Lee H, Kakuta T, Ye JC, Jang IK. A novel deep learning model for a computed tomography diagnosis of coronary plaque erosion. Sci Rep. 2023 Dec 27;13(1):22992. doi: 10.1038/s41598-023-50483-9. PMID 38151502
- [Derived] Suzuki K, Niida T, Yuki H, Kinoshita D, Fujimoto D, Lee H, McNulty I, Takano M, Nakamura S, Kakuta T, Mizuno K, Jang IK. Coronary Plaque Characteristics and Underlying Mechanism of Acute Coronary Syndromes in Different Age Groups of Patients With Diabetes. J Am Heart Assoc. 2023 Dec 5;12(23):e031474. doi: 10.1161/JAHA.123.031474. Epub 2023 Nov 28. PMID 38014673
- [Derived] Kinoshita D, Suzuki K, Usui E, Hada M, Yuki H, Niida T, Minami Y, Lee H, McNulty I, Ako J, Ferencik M, Kakuta T, Jang IK. High-Risk Plaques on Coronary Computed Tomography Angiography: Correlation With Optical Coherence Tomography. JACC Cardiovasc Imaging. 2024 Apr;17(4):382-391. doi: 10.1016/j.jcmg.2023.08.005. Epub 2023 Sep 13. PMID 37715773
- [Derived] Seegers LM, DeFaria Yeh D, Yonetsu T, Sugiyama T, Minami Y, Soeda T, Araki M, Nakajima A, Yuki H, Kinoshita D, Suzuki K, Niida T, Lee H, McNulty I, Nakamura S, Kakuta T, Fuster V, Jang IK. Sex Differences in Coronary Atherosclerotic Phenotype and Healing Pattern on Optical Coherence Tomography Imaging. Circ Cardiovasc Imaging. 2023 Aug;16(8):e015227. doi: 10.1161/CIRCIMAGING.123.015227. Epub 2023 Jul 28. PMID 37503629
- [Derived] Yuki H, Sugiyama T, Suzuki K, Kinoshita D, Niida T, Nakajima A, Araki M, Dey D, Lee H, McNulty I, Nakamura S, Kakuta T, Jang IK. Coronary Inflammation and Plaque Vulnerability: A Coronary Computed Tomography and Optical Coherence Tomography Study. Circ Cardiovasc Imaging. 2023 Mar;16(3):e014959. doi: 10.1161/CIRCIMAGING.122.014959. Epub 2023 Mar 3. PMID 36866660
- [Derived] Araki M, Sugiyama T, Nakajima A, Yonetsu T, Seegers LM, Dey D, Lee H, McNulty I, Yasui Y, Teng Y, Nagamine T, Kakuta T, Jang IK. Level of Vascular Inflammation Is Higher in Acute Coronary Syndromes Compared with Chronic Coronary Disease. Circ Cardiovasc Imaging. 2022 Nov;15(11):e014191. doi: 10.1161/CIRCIMAGING.122.014191. Epub 2022 Nov 3. PMID 36325895
- [Derived] Nakajima A, Sugiyama T, Araki M, Seegers LM, Dey D, McNulty I, Lee H, Yonetsu T, Yasui Y, Teng Y, Nagamine T, Nakamura S, Achenbach S, Kakuta T, Jang IK. Plaque Rupture, Compared With Plaque Erosion, Is Associated With a Higher Level of Pancoronary Inflammation. JACC Cardiovasc Imaging. 2022 May;15(5):828-839. doi: 10.1016/j.jcmg.2021.10.014. Epub 2021 Nov 8. PMID 34876381